CLINICAL TRIAL: NCT03166657
Title: Role of Office Hysteroscopy in Cases of Secondary Infertility After Cesarean Section
Brief Title: Office Hysteroscopy in Secondary Infertility After Cesarean Section
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Ahmad Abdelraof Ahmad Askar, principal investigator, Assiut University
Other Study IDs: OHCS
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: office hysteroscopy — A speculum is first inserted into the vagina. The hysteroscope is then inserted and gently moved through the cervix into uterus. Carbon dioxide gas or a fluid, such as saline will be put through the hysteroscope into uterus to expand it. The gas or fluid helps see the lining more clearly. The amount of fluid used is carefully checked throughout the procedure

SUMMARY:
All women with history of secondary infertility after caesarean section will be subjected to office hysteroscopy according to Royal college of obstetrics and gynecology guidelines to diagnose any subtle uterine abnormalities not detected by conventional means.

Hysteroscopic examination will be done during the proliferation phase of the menstrual cycle.

The hysteroscopic evaluation will include assessment of the cervical canal, intrauterine lesions, the endometrium and the uterotubal junction. .

If hysteroscopy reveal a lesion, its type, size, location will be recorded. Transvaginal ultrasound will be done after the procedure to detect fluid in the douglas pouch to confirm patent tubes.

Asses the uterine scar in details.

ELIGIBILITY:
Inclusion Criteria:

* Patients with secondary infertility more than 2 years after cesarean section.
* Normal semen analysis
* Normal hysterosalpingography or laparoscopy within 1year
* Evidence of ovulation by transvaginal ultrasound

Exclusion Criteria:

* • Cases with abnormal semen parameters.

  * Patients with abnormal hysterosalpingography.
  * Patients with anovulation.
  * Hormonal disturbances; high level of prolactin, thyroid hormone disturbances, very high or very low follicular stimulating hormone and luteinizing hormone
  * Patients known to be epileptic or with history of fits.
  * Cardiac patients ( valve diseases, ischemic, arrhythmic)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include all secondary infertile cases after cesarean section who presented to infertility clinic at Women health Hospital, Assiut University
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
percentage of patients with abnormal scar findings in hysteroscopy | 1 year
  color of the scar and presence of niche

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boivin J, Bunting L, Collins JA, Nygren KG. International estimates of infertility prevalence and treatment-seeking: potential need and demand for infertility medical care. Hum Reprod. 2007 Jun;22(6):1506-12. doi: 10.1093/humrep/dem046. Epub 2007 Mar 21. PMID 17376819
- [Background] Collins JA, Crosignani PG. Unexplained infertility: a review of diagnosis, prognosis, treatment efficacy and management. Int J Gynaecol Obstet. 1992 Dec;39(4):267-75. doi: 10.1016/0020-7292(92)90257-j. PMID 1361459